CLINICAL TRIAL: NCT02201147
Title: Prospective Comparison of Cold Snare Polypectomy and Cold Forceps Polypectomy Using Narrow-band Imaging Endoscopy for Diminutive Colorectal Polyps
Brief Title: Cold Snare Polypectomy Vs. Cold Forceps Polypectomy Using Narrow-band Imaging Endoscopy for Removal of Diminutive Colorectal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Soo-kyung Park, Clinical assistant professor, Soonchunhyang University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2014-04-041
Record Dates: First submitted 2014-07-22; First posted 2014-07-25 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Polyp of Large Intestine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cold biopsy polypectomy (Experimental)
  Interventions: Procedure: Cold biopsy polypectomy; Device: Cold biopsy polypectomy
- Cold snare polypectomy (Experimental)
  Interventions: Procedure: Cold snare polypectomy; Device: Cold snare polypectomy

INTERVENTIONS:
Procedure: Cold biopsy polypectomy — removal of eligible polyps using cold biopsy technique until no polyp was visible by narrow-band imaging endoscopy
  Arms: cold biopsy polypectomy
Procedure: Cold snare polypectomy — removal of eligible polyps using cold snare polypectomy technique
  Arms: Cold snare polypectomy
Device: Cold snare polypectomy — mini (10 mm open diameter) size electrosurgical snare without application of electrocautery
  Arms: Cold snare polypectomy
Device: Cold biopsy polypectomy — standard- capacity forceps with narrow band imaging endoscopy
  Arms: cold biopsy polypectomy

SUMMARY:
The purpose of this study is to compare cold snare polypectomy and cold forceps polypectomy using narrow-band imaging endoscopy for removal of diminutive colorectal polyps.

DETAILED DESCRIPTION:
Previous study found Cold snare polypectomy a preferable technique in comparison to cold biopsy for diminutive polyps when assessed for completeness of resection. However, it is expected that cold biopsy polypectomy with advanced endoscopy, such as chromoendoscopy or narrow-band imaging endoscopy, increase completeness of resection. One study showed 90% of the diminutive polyps were completely resected using cold biopsy polypectomy with chromoendoscopy. However, no study compared cold snare polypectomy and cold biopsy polypectomy using Narrow-band Imaging endoscopy for Removal of Diminutive Colorectal Polyps.

The aim of this study is to compare cold snare polypectomy and Cold biopsy Polypectomy Using Narrow-band Imaging Endoscopy for Removal of Diminutive Colorectal Polyps

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of 20 years undergoing routine colonoscopy (screening, surveillance, or diagnostic)

Exclusion Criteria:

* patients taking antiplatelet or anticoagulant therapy during the past 1 week of the procedure
* known coagulopathy
* history of inflammatory bowel diseases
* American Society of Anesthesiology class III or more
* pregnancy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2014-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
complete histologic polyp eradication rate | 2 weeks

SECONDARY OUTCOMES:
rates of tissue retrieval per polyp | 2 weeks

OTHER OUTCOMES:
polypectomy procedure times | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bong Min Ko, MD, Principal Investigator — SoonChunHyang University School of Medicine
Locations (1):
- Soonchunhyang University Hospital, Bucheon, Bucheon-si, South Korea

REFERENCES:
- [Derived] Park SK, Ko BM, Han JP, Hong SJ, Lee MS. A prospective randomized comparative study of cold forceps polypectomy by using narrow-band imaging endoscopy versus cold snare polypectomy in patients with diminutive colorectal polyps. Gastrointest Endosc. 2016 Mar;83(3):527-32.e1. doi: 10.1016/j.gie.2015.08.053. Epub 2015 Sep 7. PMID 26358331